CLINICAL TRIAL: NCT01168258
Title: Evaluation of Single Nucleotide Polymorphisms (SNPs) in Patients With and Without Diabetic Macular Edema
Status: Terminated | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100169; 10-EI-0169
Record Dates: First submitted 2010-07-22; First posted 2010-07-23 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2013-08-07

CONDITIONS: Diabetic Retinopathy; Diabetic Macular Edema
Keywords: Diabetic Retinopathy; Diabetes; Single Nucleotide Polymorphism (SNP); Diabetic Macular Edema
MeSH Terms: conditions — Diabetic Retinopathy; Diabetes Mellitus

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- Diabetic macular edema (DME) is a common condition in people with diabetes. DME occurs when blood vessels in the eye leak fluid, resulting in swelling inside the back of the eye and progressive vision loss. Research has shown that good blood sugar control can reduce the risk and severity of DME. However, not all diabetic patients with poor blood sugar control develop DME, and some patients develop DME despite excellent blood sugar control. This suggests that other factors, such as genes or inherited traits, may predispose or protect a diabetic patient from developing DME.

Objectives:

- To investigate genetic factors that may influence the development of diabetic macular edema.

Eligibility:

- Individuals at least 18 years of age who have type 2 diabetes, with or without diabetic macular edema.

Design:

* The study will require one visit to the National Institutes of Health eye clinic.
* Participants will be screened with a medical history and basic eye examination. Individuals who have certain eye diseases other than DME may not be allowed to enroll in the study.
* Participants will provide a blood sample, and will receive fluorescein angiography (an injection of fluorescein dye, after which a camera will take pictures of the dye as it flows through the blood vessels in the eye).
* No treatment will be provided as part of this protocol.

DETAILED DESCRIPTION:
Objective:

The objective of this study is to test the hypothesis that genetic polymorphisms of vascular endothelial growth factor (VEGF), erythropoietin (EPO), endothelin-1 (EDN1) and receptor for advanced glycation end product (RAGE) genes are associated with the development of diabetic macular edema (DME).

Study Population:

Two hundred case participants with DME and 200 diabetic controls without DME will be enrolled.

Design:

This is a longitudinal, genetic association study evaluating whether single nucleotide polymorphisms (SNPs) in VEGF, EPO, EDN1 and RAGE genes affect the development and progression of DME. All participants will provide a blood sample, undergo an eye examination, optical coherence tomography (OCT) and fluorescein angiography (FA) and discuss their medical, family and social history. Case participants with DME and diabetic control participants without DME will be allowed to receive standard-of-care treatment at the NEI under this protocol.

Outcome Measures:

The primary outcome variable is the genotype frequency of SNPs in the above specific genes of DME and control participants. Secondary outcomes are serum levels of VEGF, EPO, EDN1 and AGE, plasma biomarkers such as mRNA and ophthalmic measurements (visual acuity and imaging results such as FA and OCT results). The longitudinal outcome measure includes investigating associations between the studied genetic polymorphisms and the long-term response to standard-of-care therapy.

ELIGIBILITY:
* INCLUSION CRITERIA:

All participants must meet the following criteria:

Participant is diagnosed with type 2 diabetes prior to enrollment.

Participant must understand and sign this protocol s informed consent document and agree to provide a blood sample for analysis.

Participant must be 18 years of age or older.<TAB>

DME Participants (cases):

Participant is diagnosed with active DME defined by fluorescein leakage associated with either central retinal thickness greater than 260 microns on spectral domain OCT or cystic changes present on OCT.

OR

Participant has evidence of focal laser scars indicative of prior DME Investigators will verify the laser therapy was performed for DME via medical records, fluorescein angiograms or photographs.

Non-DME Participants (controls)

Participant has no evidence of DME defined fluorescein leakage associated with either central retinal thickness greater than 260 microns on spectral domain OCT or cystic changes present on OCT.

Participant has no evidence of focal laser scars indicative of prior DME.

EXCLUSION CRITERIA:

Participant has another retinal disease that may confound the evaluation of the DME. Examples include vein occlusions, uveitic macular edema or neovascular age-related macular degeneration.

Participant has opacities of the ocular media, limitations of pupillary dilation or other problems sufficient to preclude adequate dilated examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2010-07-07; Study Completion 2013-08-07

PRIMARY OUTCOMES:
Genotype frequency of SNP in the study genes of DME participants and control participants.

SECONDARY OUTCOMES:
Secondary outcomes are ophthalmic measurements, including visual acuity, FA and OCT data, to investigate associations between detected genetic polymorphisms and response to conventional diabetic retinopathy treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Meyerle, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Wild S, Roglic G, Green A, Sicree R, King H. Global prevalence of diabetes: estimates for the year 2000 and projections for 2030. Diabetes Care. 2004 May;27(5):1047-53. doi: 10.2337/diacare.27.5.1047. PMID 15111519
- [Background] Risch NJ. Searching for genetic determinants in the new millennium. Nature. 2000 Jun 15;405(6788):847-56. doi: 10.1038/35015718. PMID 10866211
- [Background] Martin ER, Lai EH, Gilbert JR, Rogala AR, Afshari AJ, Riley J, Finch KL, Stevens JF, Livak KJ, Slotterbeck BD, Slifer SH, Warren LL, Conneally PM, Schmechel DE, Purvis I, Pericak-Vance MA, Roses AD, Vance JM. SNPing away at complex diseases: analysis of single-nucleotide polymorphisms around APOE in Alzheimer disease. Am J Hum Genet. 2000 Aug;67(2):383-94. doi: 10.1086/303003. Epub 2000 Jun 21. PMID 10869235